CLINICAL TRIAL: NCT00786799
Title: A Randomized, Double-Blind, Placebo-Controlled 12-week Study to Investigate the Effect of Omega-3 Fatty Acids on Hyperactivity in Childhood Autism
Brief Title: Omega-3 Fatty Acids for Autism Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Autism Speaks (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 200816175-1
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Results first posted 2012-08-31 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-07

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder | interventions — Fatty Acids, Omega-3; Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omega-3 Fatty Acids (Active Comparator)
  Interventions: Dietary Supplement: Omega-3 Fatty Acids
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Omega-3 Fatty Acids

INTERVENTIONS:
Dietary Supplement: Omega-3 Fatty Acids — Omega-3's are administered in the form of an orange pudding made by Coromega
  1 mg of omega-3 fatty acid 2 times per day
  Other Names: Omega-3, N-3 Fatty Acid
  Arms: Omega-3 Fatty Acids
Dietary Supplement: Omega-3 Fatty Acids — Omega-3 Fatty Acids in orange pudding form
  1 packet two times per day
  Other Names: Omega-3, N-3 Fatty Acid
  Arms: Placebo

SUMMARY:
Omega-3 fatty acids are among the most commonly used CAM (Complementary Alternative Medical) therapies, and have been reported to be currently used by 28.7% of children with autism. Two published case series noted that families reported large improvements in the core feature of autism when children were given omega-3 fatty acids. Low levels of omega-3 fatty acids have been noted in children with autism, which suggests normalizing the omega-3 fatty acid levels could produce improvements in the symptoms seen in many children with autism.

This study is a 12-week randomized, double blind, placebo-controlled clinical trial for 24 male and female children aged 3 to 8 years with autism. Patients who are currently using omega-3 would need to discontinue omega-3 fatty acids for 8 weeks before they are able to participate in the study. All study participants who meet all inclusion and no exclusion criteria at the initial screening visit and sign the consent form will then complete baseline assessments of the outcome measures (validated instruments of hyperactivity, communication, social interaction, and behavior) and be randomly assigned to 12 weeks of omega-3 fatty acids at a dose of 1 gm per day or an identical placebo. The child's behavior will be measured and evaluated at the MIND Institute at the beginning of the study and at study closing. All study families will come in for a follow-up visit at weeks 4 and 8 to assess medication compliance and side effects to study medication.

After 12 weeks of treatment, all outcome measures including laboratory tests and side effect profiles will be repeated. All patients who complete the study will receive a 12-week supply of omega-3. This would also provide patients who were on placebo with active medication. No follow-up visits are needed once the patient finishes the double-blind portion of the study.

DETAILED DESCRIPTION:
Clinical measures will be used to assess diagnosis and efficacy. All clinical assessments will take place at the M.I.N.D. Institute. Baseline and termination measures will include the Aberrant Behavior Checklist (ABC), Peabody Picture Vocabulary Test (PPVT-III), Expressive Vocabulary Test (EVT), Social Responsiveness Scale (SRS), Behavior Assessment System for Children (BASC), and Clinical Global Impression Improvement (CGI-I). The, the Wechsler Preschool Primary Scale of Intelligence - Revised (WPPSI-R), the Wechsler Intelligence Scale for Children (WISC) or the Stanford-Binet will be administered to measure IQ.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of autism as defined by DSM-IV TR and scores above the cutoff on the Autism Diagnostic Observation Scale (ADOS) and the Social Communication Questionnaire (SCQ)
* Age three to eight years
* Non-verbal IQ of 50 or above
* Children on a stable medical regimen for the past 2 months and no plans to change medical therapy for the study period

Exclusion Criteria:

* Individuals with allergy or hypersensitivity to fish or nuts
* Diabetes
* Bleeding disorder, current use of anticoagulant or anti-platelet therapy, or recent surgery
* Clinical evidence of seizure disorder
* Cancer
* Fragile X or other known genetic cause of autism
* Perinatal brain injury
* Evidence for malnutrition seen in abnormal albumin level
* Other serious medical illness
* Current use of omega-3 fatty acids

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2008-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Bent, MD, Principal Investigator — University of California, San Francisco; Robert L Hendren, DO, Principal Investigator — UC San Francisco
Locations (1):
- UC San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] Lunsky Y, P Hastings R, Weiss JA, M Palucka A, Hutton S, White K. Comparative Effects of Mindfulness and Support and Information Group Interventions for Parents of Adults with Autism Spectrum Disorder and Other Developmental Disabilities. J Autism Dev Disord. 2017 Jun;47(6):1769-1779. doi: 10.1007/s10803-017-3099-z. PMID 28374207
- [Derived] Bent S, Bertoglio K, Ashwood P, Bostrom A, Hendren RL. A pilot randomized controlled trial of omega-3 fatty acids for autism spectrum disorder. J Autism Dev Disord. 2011 May;41(5):545-54. doi: 10.1007/s10803-010-1078-8. PMID 20683766

RESULTS

PARTICIPANT FLOW:
Groups:
- Omega-3 Fatty Acids: Omega-3 fatty acids were provided as orange-flavored pudding packets (Coromega®, Vista, CA) containing 650 mg of omega-3 fatty acids, including 350 mg of eicosapentanoic acid (EPA) and 230 mg of docosahexanoic acid (DHA), given twice daily for a daily dose of 1.3 g of omega-3 fatty acids (and 1.1 g of DHA + EPA).
- Placebo: Placebo packets had the same orange-flavored pudding with an identical appearance and taste, but included safflower oil instead of the fish oil (omega-3 fatty acids). Safflower oil was used because it is has a similar texture and is comprised of fatty acids (but not omega-3 fatty acids), and this allowed for an examination of the unique of effects of omega-3 fatty acids compared to "non-omega-3" fatty acids.
Period: Overall Study
Arm/Group | Omega-3 Fatty Acids | Placebo
Started | 14 | 13
Completed | 13 | 12
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omega-3 Fatty Acids | Placebo | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 13 | 27
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 5.85 (1.83) | 5.82 (1.42) | 5.83 (1.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 13 | 11 | 24
Region of Enrollment [Number; unit: participants]
  United States | 14 | 13 | 27

OUTCOME MEASURES:

1. Primary Outcome: Group-specific and Comparison of Change in Aberrant Behavior Checklist-Hyperactivity Subscale Score (Active Omega-3 Group Only, Placebo Group Only and Comparison Between Groups)
Description: Hyperactivity subscale of Aberrant Behavior checklist (ABC-H): measure of assessing changes in symptoms of hyperactivity in children with autism (survey that was normed on a developmentally delayed population of children and adults and is usually completed by a parent or caregiver. Items are rated on a 4-point scale from "no problem" to "major problem"). ABC-H Subscale Score ranges from 0 (best) to 45 (worst). A negative change signifies improvement.
Time Frame: Baseline and 1 year
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Active Omega-3: Mean and Standard Deviation of Change in Aberrant Behavior Checklist-Hyperactivity Subscale Score within Omega-3 Group Only
- Placebo: Mean and Standard Deviation of Change in Aberrant Behavior Checklist-Hyperactivity Subscale Score within Placebo Group Only
- Comparison Between Omega-3 and Placebo Groups: Comparison of Change in Aberrant Behavior Checklist-Hyperactivity Subscale Score between Omega-3 and Placebo groups (p-value given in statistical analysis section)
Arm/Group | Active Omega-3 | Placebo | Comparison Between Omega-3 and Placebo Groups
Number analyzed (Participants) | 13 | 12 | 25
scores on a scale | 2.7 (4.8) | 0.3 (7.2) | 2.3 (6.1)
Statistical Analysis 1: Comparison: Comparison Between Omega-3 and Placebo Groups; The null hypothesis is that the mean change in Aberrant Behavior Checklist Hyperactivity subscale (ABC-H) score is the same for both groups; Test type: Superiority or Other; p = 0.40, t-test, 2 sided; Mean Difference (Net) = 2.3, Standard Deviation 6.1

2. Secondary Outcome: Change in Percentage of Serum Omega-3 Fatty Acids
Description: Change in percentage calculated as (100% * ((One Year - Baseline)/Baseline)
Time Frame: Baseline and 1 year
Measure: Mean (Standard Deviation); unit: Percent change of levels of fatty acid
Groups:
- Active Omega-3 Group: Change in Levels of Omega 3 Fatty Acids: Change in percentage of serum levels of Omega-3 fatty acids in the active Omega-3 group (100% * ((One Year - Baseline)/Baseline)
- Placebo Group: Change in Levels of Omega 3 Fatty Acids: Change in percentage of serum levels of Omega-3 fatty acids in the placebo group (100% * ((One Year - Baseline)/Baseline).
Arm/Group | Active Omega-3 Group: Change in Levels of Omega 3 Fatty Acids | Placebo Group: Change in Levels of Omega 3 Fatty Acids
Number analyzed (Participants) | 13 | 12
Percent change of levels of fatty acid | 2.54 (2.8) | -0.10 (0.3)

3. Secondary Outcome: Change in Serum TNFα (Cytokine) Level
Time Frame: Baseline and 1 year
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Active Omega-3 Group: Change in TNFα | Placebo Group: Change in TNFα
Number analyzed (Participants) | 13 | 12
pg/ml | 1.3 (2.5) | -0.9 (2.1)

ADVERSE EVENTS:
Arm/Group | Omega-3 Fatty Acids | Placebo
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 5/14 | 4/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omega-3 Fatty Acids (N=14) | Placebo (N=13)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nose Bleed (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
GI Symptoms (Gastrointestinal disorders) | 1 (1) | 0 (0)
Increased Hyperactivity (Nervous system disorders) | 0 (0) | 3 (3)
Increased Self-Stimulating Behavior (Nervous system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
1. Small sample size which results in a limited power to detect small to moderate treatment effects.
2. Relatively mild level of hyperactivity in both groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No